CLINICAL TRIAL: NCT04628611
Title: Comparison Between Rigid Video Assisted Laryngoscopy vs Flexible Laryngoscopy in Anticipated Difficult Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IORG000381
Record Dates: First submitted 2020-10-15; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Intubation
Keywords: video laryngoscopy; Flexible intubating bronchoscope; Anticipated difficult intubation

STUDY DESIGN:
Intervention Model Description: two equal groups; group (V) using video laryngoscope(53) and group (F) using flexible intubating laryngoscopy(53).
Who Masked: Participant
Masking Description: the participant does not know which group the patient belongs to as every patient was consented for both devices which were ready in the operating theatre
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video laryngoscopy Group (V) using Storz c-mac laryngoscope (Active Comparator): video laryngoscope without a channel used for endotracheal intubation, the device used to obtain a view of the larynx, and the endotracheal tube is passed through the vocal cords independent of the device. The device is connected to the monitor via connecting cable
  Interventions: Device: Video laryngoscopy
- The flexible intubating laryngoscopy Group (F) using Storz flexible intubation video endoscope set (Active Comparator): The flexible intubating scope is used to locate the vocal cords and acts as a stylet for the endotracheal tube once the scope is placed into the trachea.This device consists of a flexible insertion cord that contains a small camera at the tip, used to transmit images to camera head. The cord includes a channel for a light source, a working channel for suction or administration of oxygen or local anesthetic, and a cable that allows the operator to flex the tip of the scope. The cord attaches to a handle with a light source,camera head control lever for flexion/extension of the tip, and a working channel port. The device is connected to the monitor via connecting table
  Interventions: Device: Flexible intubating laryngoscopy

INTERVENTIONS:
Device: Video laryngoscopy — Endotracheal intubation using video laryngoscopy
  Other Names: Storz c-mac laryngoscopy
  Arms: Video laryngoscopy Group (V) using Storz c-mac laryngoscope
Device: Flexible intubating laryngoscopy — Endotracheal intubation using flexible intubating laryngoscope
  Other Names: Storz flexible intubation video endoscope set
  Arms: The flexible intubating laryngoscopy Group (F) using Storz flexible intubation video endoscope set

SUMMARY:
This is a randomized control study where adult patients had been divided randomly into two equal groups using video laryngoscope in group (V) and flexible intubating laryngoscope in group (F)

DETAILED DESCRIPTION:
Routine pre-operative assessment including history taking, clinical examination, and laboratory tests. Patients were admitted to the operating room with a small 20G IV cannula after applying inclusion & exclusion criteria and airway assessment by applying El Ganzuri multivariate risk index for difficult intubation which include assessment of the following : inter-incisor gap, Mallampati classification, head &neck movement, buck teeth prognathism, thyromental distance, body weight and history of difficult intubation.

Operating room was prepared using :

Difficult airway cart that includes different size oral airways, endotracheal tubes, different sizes face masks & laryngeal airway masks Suction apparatus to be ready for use Video laryngoscopy The flexible intubating laryngoscopy with the tube mounted over the fiberscope before the procedure.

Standard monitoring devices were applied including ECG, non invasive blood pressure. pulse oximetry and capnography after intubation Patients were then pre-oxygenated via face mask for three minutes and using 0.01 mic/kg atropine then general anesthesia is induced using fentanyl 1-2 mic/kg followed by propofol 2 mg/kg and esmeron 0.5 mg/kg.

The patient is mechanically ventilated using face mask until full relaxation is established after 3-5 minutes. The intubation is done using video laryngoscope in group (v) or using flexible intubating laryngoscopy in group (f) In the first group (v) The video laryngoscope was introduced with the patient appropriately positioned, the operator used the left hand to introduce the video laryngoscope into the midline of the Oropharynx and gently advances until the blade tip pass the posterior portion of the tongue. Using video visualization, the ETT was then advanced on a smooth curve through the glottis and intubation proceeds. Viewing the entire insertion step on the video screen allows the operator to quickly become facile with the motion of gently rotating or angling the tube using the right hand to redirect as necessary.

In the second group(f) patients positioned supine with the operator standing at the head of the bed. Simple chin lift and jaw thrust may improve the view through the flexible laryngoscopy and also help to prevent airway obstruction. The endotracheal tube should be lubricant to facilitate its subsequent advancement into the trachea. Once the endotracheal tube is in place, the scope is removed, and the patient is ventilated. Flexible intubating laryngoscopy is often performed with the operator looking through the eyepiece. However, connecting the flexible laryngoscopy to a monitor is often advantageous.

After collecting demographic data of the patient (age, sex, body mass index & ASA) The following parameters will be measured :

Intubation time, Hemodynamic parameters, success rate and number of attempts & incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

1. El-Ganzouri score: 2, 3, 4 (Table 1)
2. American Society of Anesthesiology (ASA) I, II, III
3. Elective surgeries

Exclusion Criteria:

1. Refusal of participation
2. Patients who need a surgical airway (e.g. patients with highly obstructing laryngeal lesions such as cancer tongue, larynx& maxilla).
3. Patients with laryngeal trauma, especially in those with suspected cricotracheal separation.
4. Patients with craniofacial trauma.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Intubation time | Through study completion (Assessment done at the same time of doing intubation) within 60 seconds
  time from initiation of intubation (application of the laryngoscope into mouth) to ETCO2 detection from the ETT. In cases with failed intubation it was considered from initiationof intubation till failure. Measured by seconds

SECONDARY OUTCOMES:
Heart rate | At the same time of doing the intubation within 15 minutes
  Measured by(beat/ minute). measured during baseline (just before induction of anesthesia), 3 minutes & 10 minutes after intubation.
Number of attempts | AT the same time of doing the intubation within 30 minutes
  Airway instrumentation will be interrupted if oxygen saturation decreases below 92% and patients are ventilated via a face mask. After 3 failed trials the procedure is considered unsuccessful with insertion of classical LMA of appropriate size, correct placement should be confirmed by capnography, manual ventilation with 100% oxygen should be done and awaken the patient
Incidence of complications | From time of intubation till end of surgery and extubation within 10 hours
  sore throat, mucosal or pharyngeal injury, and esophageal intubation, marked desaturation and unsatisfactory blood gases
Blood pressure | At the same time of intubation within 15 minutes
  Measured by mm/Hg measured during baseline (just before induction of anesthesia), 3 minutes & 10 minutes after intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Essam AH Mahran, MD, Study Director — Assistant Professor of Anesthesia, ICU, and Pain Management, NCI, Cairo